CLINICAL TRIAL: NCT06910345
Title: Effect of Melatonin Patches on Sleep Quality in Patients Undergoing Urological Surgery
Brief Title: Effect of Melatonin Patches on Sleep in Urological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Cagla Toprak, Dr., Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09/06 number, 19.11.2024
Record Dates: First submitted 2025-03-25; First posted 2025-04-04 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2024-12

CONDITIONS: Urological Surgery
Keywords: transdermal melatonin,; urological surgery; sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin group (Experimental): Before the patient goes to sleep, the nurse will ensure that the room is quiet and dark, as exposure to light suppresses melatonin. First, the introductory characteristics form and the Richard's-Campbel Sleep Scale will be completed for patients assigned to the melatonin group. Melatonin patches will be placed by a nurse not involved in the study at 8:00 PM before going to sleep (on the upper chest or forearm, as determined by the patient). The patches will remain on for an average of 6-10 hours, depending on the patient's preferred sleep hygiene. If a patient wishes to have the patch removed during the night, they will be instructed to ask the clinic nurse to do this. The Richard's-Campbel Sleep Scale will be completed when the patient is fully awake after the melatonin patch is removed one hour before the patient goes to the operating room on the morning of the surgery.
  Interventions: Other: A skin patch (2.1 mg melatonin) was applied to the melatonin group. The melatonin patches will be placed at 8:00 PM (on the upper chest or forearm, as determined by the patient) before going to sleep
- control group (No Intervention): Patients in the control group will not undergo any intervention other than the standard care protocol.

INTERVENTIONS:
Other: A skin patch (2.1 mg melatonin) was applied to the melatonin group. The melatonin patches will be placed at 8:00 PM (on the upper chest or forearm, as determined by the patient) before going to sleep — A skin patch (2.1 mg melatonin) was applied to the melatonin group.
  Arms: Melatonin group

SUMMARY:
Patients undergoing urological surgery may experience a decrease in sleep quality due to many factors such as hospitalization, different environment, pain, stress and anesthesia. After surgery, melatonin secretion decreases and circadian rhythm becomes irregular in patients. This problem can lead to sleep disorders in patients. Melatonin is an important hormone that regulates both sleep and circadian rhythms. The aim of this study is to observe the effect of a melatonin skin patch designed to produce melatonin in a way that ensures a stable increase in melatonin levels in the blood, on patients undergoing urological surgery.

DETAILED DESCRIPTION:
The purpose of this study was to observe the effect of a melatonin skin patch designed to produce melatonin, which would provide a stable increase in blood melatonin levels, on patients undergoing urological surgery. The patients were applied a melatonin patch before surgery. The other group received routine nursing care.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone planned urological surgery,

  * Those who receive melatonin patch therapy,
  * Those who are between the ages of 18-70,
  * Those whose hemodynamic conditions are stable will be included.

Exclusion Criteria:

* •Patients who used different sleeping pills/hypnotics during the study period,

  * Patients with delirium/psychiatric illness,
  * Patients with hearing and speech problems will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
sleep quality | The Richards-Campbell Sleep Scale will be completed at 20:00 the evening before surgery and at 06:00 the morning of surgery.
  Sleep is examined in the parameter and scored between 100 'very suitable' and 0 'not suitable'. The higher the score obtained from the scale, the higher the patient's sleep quality is considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Atlas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: April 15, 2025

REFERENCES:
- [Result] Aeschbach D, Lockyer BJ, Dijk DJ, Lockley SW, Nuwayser ES, Nichols LD, Czeisler CA. Use of transdermal melatonin delivery to improve sleep maintenance during daytime. Clin Pharmacol Ther. 2009 Oct;86(4):378-82. doi: 10.1038/clpt.2009.109. Epub 2009 Jul 15. PMID 19606092